CLINICAL TRIAL: NCT05860686
Title: Does Post-operative Rinsing With a Monoject Syringe Result in as Much Post-operative Pain After Surgical Removal of Lower Impact Third Molars as no Post-operative Rinsing: a Randomized Controlled Equivalence Trial
Acronym: RITOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Jeroen van der Sleen, Oral an Maxillo facial surgeon, Isala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL81366.075.22
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Third Molar

STUDY DESIGN:
Intervention Model Description: Double blind randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No rinsing (Active Comparator)
  Interventions: Other: Monoject syringe
- Monoject rinsing (Experimental)
  Interventions: Other: Monoject syringe

INTERVENTIONS:
Other: Monoject syringe — monoject syringe is used to clean the wound

SUMMARY:
Many authors have advocated different methods of treating alveolar osteitis. Despite many years of research, however, little progress has been made and so a study with large enough sample and standard outcome measures is warranted.

Goal of this study is assess the effect of postoperative use of a monoject syringe on postoperative complaints after surgical removal of a lower third molar.

DETAILED DESCRIPTION:
One of the most common postoperative complications after the removal of a third molar is a condition known as dry socket. This term has been in use since 1896. Since then several other terms have been used, including alveolar osteitis, postoperative alveolitis, alveolitis, sicca dolorosa and fibriniolytic alveolitis. Bim labelled the complication fibrinolytic alveolitis which is the most accurate of the terms, but also the least used. The condition has generally been characterised by delayed healing associated with degradadtion of clot, and is usually accompanied by persistent, radiating, pain postoperativively in and around the extraction site that is not easily relieved by analgesics. Because of the pain, swelling and trismus, patients also tend to have a greater need for painkillers. If it is possible to reduce the amount and severity of postoperative pain felt by patients the postoperative period would be more endurable, the quality of life will be less affected, and in addition to this it is possible that the amount of analgesics taken by patients after surgery could be lowered7. It can be a burden for both patients an surgeons and my result in a loss of productivity because at least 45% of patients require multiple visits to the surgeon.

Objective of the study:

Many authors have advocated different methods of treating alveolar osteitis. Despite many years of research, however, little progress has been made and so a study with large enough sample and standard outcome measures is warranted.

Goal of this study is assess the effect of postoperative use of a monoject syringe on postoperative complaints after surgical removal of a lower third molar

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria: patients over 18 years of age (non-smoking) referred for removal of a wisdom tooth in the mandible. Patient has ASA I.

Exclusion Criteria:

* Patient is younger than 18 years

Patient has an ASA of II,III en IV

Patient has only one maxillary third molar that needs to be extracted/removed

Patient has an active pericoronitis

In case of planned coronectomy

Patient has trismus

Patient has chronic pain

Patient is pregnant

Patient has a known allergy for ibuprofen of other NSAID's

Patient has a known allergy for articaine of epinefrine

Intra-operative compilations for example excessive bleeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
NRS pain | 7 days after treatment
  pain score

IPD SHARING:
Plan to Share IPD: Undecided